CLINICAL TRIAL: NCT00659880
Title: Clinical Application of BioCleanse Meniscus Registry
Brief Title: Clinical Application of BioCleanse Meniscus
Acronym: Meniscus
Status: Completed | Type: Observational
Sponsor: RTI Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: BioMen
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-04

CONDITIONS: Tear of Meniscus of Knee
Keywords: Meniscus transplant; Meniscal allograft; MAT; Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: BioCleanse Meniscus — Subjects will undergo routine meniscal allograft transplant surgery.

SUMMARY:
This study will follow patients after routine surgery of a meniscal allograft transplant.

DETAILED DESCRIPTION:
The BioCleanse meniscus is available to to all orthopedic surgeons for transplantation. The purpose of this registry is to allow close monitoring of a subgroup of patients receiving the BioCleanse Meniscus. All patients who have selected a BioCleanse Meniscus for their Meniscal Allograft transplant will be asked to join the registry. Outcomes will be measured by subjective subject questionnaires as well as X-rays and MRI.

ELIGIBILITY:
Inclusion Criteria:

* All patients, up to 10 who have selected a BioCleanse Meniscus transplant

Exclusion Criteria:

* Anyone not eligible for a meniscal transplant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients, between the ages of 18 and 55 years, who have selected meniscal allograft transplantation (MAT) using BioCleanse allografts will be eligible to participate in the MAT registry.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2008-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack Farr, MD, Principal Investigator — OrthoIndy -Orthopaedic Research Foundation, Inc
Locations (1):
- OrthoIndy, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Meniscal Allograft Transplant: Patients who received a BioCeanse Meniscal Allograft Transplant
Period: Overall Study
Arm/Group | Meniscal Allograft Transplant
Started | 9
6 Weeks | 9
6 Months | 9
12 Months | 7
24 Months | 6
Completed | 4 (60 months)
Not Completed | 5
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Arm/Group | Meniscal Allograft Transplant
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: The score is an index score from 0 to 100, with 0 representing extreme problems and 100 representing no problems.
Time Frame: 60 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meniscal Allograft Transplant
Number analyzed (Participants) | 4
units on a scale | 70.1 (33.6)
Statistical Analysis 1: Comparison: Meniscal Allograft Transplant; Test type: Superiority or Other; p = 0.06, Friedman

2. Secondary Outcome: MRI Assessments
Description: MRI images were assessed for integration of the meniscal allograft transplant for integration of the anterior horn, body and posterior horn.
  Images were also assessed for oedema in each of these 3 regions of the meniscus.
Time Frame: 12 months
Measure: Number; unit: participants
Groups:
- Meniscal Allograft Integration: The MRI were assessed for the integration of the posterior and anterior horns as well as the body of the meniscus.
Arm/Group | Meniscal Allograft Integration
Number analyzed (Participants) | 4
participants
  Integration of Meniscal Body | 4
  Integration of Anterior Horn | 3
  Integration of Posterior Horn | 4
  Mild Edema Anterior Horn | 2
  Mild Edema Posterior Horn | 1
  Mild Edema Meniscal Body | 0

ADVERSE EVENTS:
Time Frame: Unexpected AE data were collected at each of 5 post-operative visits: 6 weeks, 6 months, 12 months, 24 months, 60 months. All AE were documented on case report forms.
Description: Of the AE reported, 2 were definitely not related to the allograft, 2 were considered unlikely related and 2 were considered possibly related.
Arm/Group | Meniscal Allograft Transplant
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 4/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Meniscal Allograft Transplant (N=9)
Ipsilateral knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
arm fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee impinging scar (Musculoskeletal and connective tissue disorders) | 1 (1)
Chondrosis: Trochlea & Patella (Musculoskeletal and connective tissue disorders) | 1 (1)
meniscal allograft lesion (Musculoskeletal and connective tissue disorders) | 1 (1)
Contralateral (non-study) knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may present/publish in meetings, journals, theses, dissertations the results of Investigation provided that RTI will have been furnished copies of any proposed publication/presentation at least 40 days in advance of the submission. RTI will have 30 days after receipt to object & withhold consent to the proposed presentation/publication either because there is patentable subject matter which needs protection and or there is Confidential or inaccurate information contained in the publication